CLINICAL TRIAL: NCT00400335
Title: An Open Label Study to Evaluate the Impact of Novel Fixed-dose Testosterone/Dutasteride Combinations on the Relative Bioavailability of the Individual Dutasteride and Testosterone Components
Brief Title: Study On Bioavailability And Pharmacokinetics Of Various Doses Of Testosterone Administered With And Without Dutasteride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDC106222
Record Dates: First submitted 2006-11-14; First posted 2006-11-16 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Hypogonadism; Hypogonadism, Male
Keywords: Testosterone; Men; Hypogonadism; Dutasteride; DHT; Androgen deficiency
MeSH Terms: conditions — Hypogonadism; Eunuchism; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nanomilled testosterone
Drug: commercially available dutasteride
Drug: Nanomilled dutasteride
  Other Names: commercially available dutasteride; Nanomilled testosterone

SUMMARY:
The combination of testosterone and dutasteride is intended for use in hypogonadal men. This study will evaluate the bioavailability and pharmacokinetics of various doses of testosterone administered with and without dutasteride

ELIGIBILITY:
Inclusion criteria:

* Are healthy.
* Have a BMI within range of 19-32 kg/m2.
* Have not taken dutasteride for one year, or finasteride for the past 3 months.
* Have a screening PSA < 2.0ng/mL.

Exclusion criteria:

* Have had or have breast or prostate cancer, sleep apnea, psychiatric illness, or any other clinically significant current condition.
* Have a trigliceride level =500mg/dL.
* Have abnormal thyroid or hormone levels.
* Would donate more than 500 ML of blood over a 2 month period.
* Physician does not think it is a good idea for you to participate in the trial.
* Are unwilling to abstain from alcohol during the study.
* Have a positive urine drug screen test.
* Plan to change your smoking habits during the course of the trial.
* Have Hepatitis C, Hepatitis B, or HIV.
* Have a lab or ECG abnormality.
* Have high or low blood pressure.
* Have used of any investigational drug or device during the study or within 30 days prior to 1st dosing of study medication.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
lab tests for relative bioavailability of testosterone and dutasteride, | days 1, 2, 3, 19, 20, 21 & 26-31

SECONDARY OUTCOMES:
safety lab tests of various testosterone/dutasteride formulations, | days 1, 2, 3, 19, 20, 21 & 26-31.
lab tests for additional pharmacokinetic parameters for testosterone & dutasteride, | days 1, 2, 3, 19, 20, 21 & 26-31.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States